CLINICAL TRIAL: NCT05919784
Title: Examining the Effectiveness of a Group Cognitive-behavioural Treatment Program for Persistent Genital Arousal Disorder/Genitopelvic Dysesthesia
Brief Title: Examining the Effectiveness of a Group Cognitive-behavioural Treatment Program for Persistent Genital Arousal Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Caroline Pukall (Other)
Responsible Party: Sponsor-Investigator, Dr. Caroline Pukall, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 379631-3
Record Dates: First submitted 2023-06-13; First posted 2023-06-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Persistent Genital Arousal Disorder
Keywords: Persistent Genital Arousal Disorder; intervention
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive behavioural therapy (Experimental): The group therapy program (virtual, synchronous) involves elements based in Cognitive Behavioural Therapy (CBT), Acceptance and Commitment Therapy (ACT), and Dialectical Behaviour Therapy (DBT).
  Interventions: Behavioral: Cognitive behavioural therapy

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — The group therapy program (virtual, synchronous) involves elements based in Cognitive Behavioural Therapy (CBT), Acceptance and Commitment Therapy (ACT), and Dialectical Behaviour Therapy (DBT).

SUMMARY:
This study seeks to provide information regarding the effectiveness of a virtual, synchronous cognitive behavioural therapy (CBT) group program for women with Persistent Genital Arousal Disorder/Genitopelvic Dysesthesia (PGAD/GPD). The program consists of 8 weekly sessions of two hours each, which focus on education and understanding, and learning skills and strategies to manage PGAD/GPD symptoms, and related mental health and lifestyle impacts, as well as structured opportunities for discussion and shared reflection. The group therapy program involves elements based in Cognitive Behavioural Therapy (CBT), Acceptance and Commitment Therapy (ACT), and Dialectical Behaviour Therapy (DBT). Participants in the present study will provide responses to online surveys (before, during, and immediately after treatment, also 3 and 6 months after treatment) regarding their PGAD/GPD symptoms, mental health symptoms, and sexual wellness (sexual pleasure and distress).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* fluent in English
* have a physician-based diagnosis of PGAD/GPD
* reside in Ontario, Canada
* be comfortable answering questions about their health (mental and physical) and sexuality in online surveys
* be comfortable discussing their mental and physical health and PGAD/GPD symptoms in group online therapy sessions with video on

Exclusion Criteria:

* under the age of 18 years
* nonfluent in English
* lack of physician based diagnosis of PGAD/GPD
* not comfortable with answering questions about mental, physical, sexual health
* not comfortable with discussing mental and physical health and PGAD/GPD symptoms in group online therapy sessions with video on
* mental or physical health conditions that preclude involvement in group therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Anyone who self-identifies as a woman is eligible to participate.
Enrollment: 25 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Symptom intensity | Baseline
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 1 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 2 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 3 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 4 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 5 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 6 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 7 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | Week 8 of program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | 3 months after the end of the program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom intensity | 6 months after the end of the program
  Symptom intensity on a scale of 0 (no symptoms) to 10 (extremely intense symptoms). Range is 0-10. Higher scores are worse.
Symptom distress | Baseline
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 1 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 2 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 3 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 4 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 5 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 6 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 7 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | Week 8 of program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | 3 months after the end of the program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.
Symptom distress | 6 months after the end of the program
  Symptom distress on a scale of 0 (no distress) to 10 (extreme distress). Range is 0-10. Higher scores are worse.

SECONDARY OUTCOMES:
Symptom catastrophizing | Baseline
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 1 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 2 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 3 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 4 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 5 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 6 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 7 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | Week 8 of program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | 3 months after the end of the program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom catastrophizing | 6 months after the end of the program
  Pain Catastrophizing Scale, adapted to symptoms. Range is 0-52. Higher scores are worse.
Symptom self-efficacy | Baseline
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 1 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 2 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 3 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 4 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 5 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 6 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 7 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | Week 8 of program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | 3 months after the end of the program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Symptom self-efficacy | 6 months after the end of the program
  Pain Self-Efficacy Scale, adapted to symptoms. Range is 0-60. Higher scores are better.
Resilience | Baseline
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 1 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 2 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 3 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 4 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 5 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 6 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 7 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | Week 8 of program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | 3 months after the end of the program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.
Resilience | 6 months after the end of the program
  Brief Resilience Scale. Range is 6-30. Higher scores are better.

OTHER OUTCOMES:
Sexual distress | Baseline
  Sexual distress scale. Range is 0-20. Higher scores are worse.
Sexual distress | Week 4 of program
  Sexual distress scale. Range is 0-20. Higher scores are worse.
Sexual distress | Week 8 of program
  Sexual distress scale. Range is 0-20. Higher scores are worse.
Sexual distress | 3 months after the end of the program
  Sexual distress scale. Range is 0-20. Higher scores are worse.
Sexual distress | 6 months after the end of the program
  Sexual distress scale. Range is 0-20. Higher scores are worse.
Anxiety | Baseline
  Generalized Anxiety Scale. Range is 0-21. Higher scores are worse.
Anxiety | Week 4 of program
  Generalized Anxiety Scale. Range is 0-21. Higher scores are worse.
Anxiety | Week 8 of program
  Generalized Anxiety Scale. Range is 0-21. Higher scores are worse.
Anxiety | 3 months after the end of the program
  Generalized Anxiety Scale. Range is 0-21. Higher scores are worse.
Anxiety | 6 months after the end of the program
  Generalized Anxiety Scale. Range is 0-21. Higher scores are worse.
Depression | Baseline
  Patient Health Questionnaire-9. Range is 0-27. Higher scores are worse.
Depression | Week 4 of program
  Patient Health Questionnaire-9. Range is 0-27. Higher scores are worse.
Depression | Week 8 of program
  Patient Health Questionnaire-9. Range is 0-27. Higher scores are worse.
Depression | 3 months after the end of the program
  Patient Health Questionnaire-9. Range is 0-27. Higher scores are worse.
Depression | 6 months after the end of the program
  Patient Health Questionnaire-9. Range is 0-27. Higher scores are worse.
Symptom-related disability | Baseline
  Pain disability index, adapted for symptoms. Range is 0-70. Higher scores are worse.
Symptom-related disability | Week 4 of program
  Pain disability index, adapted for symptoms. Range is 0-70. Higher scores are worse.
Symptom-related disability | Week 8 of program
  Pain disability index, adapted for symptoms. Range is 0-70. Higher scores are worse.
Symptom-related disability | 3 months after the end of the program
  Pain disability index, adapted for symptoms. Range is 0-70. Higher scores are worse.
Symptom-related disability | 6 months after the end of the program
  Pain disability index, adapted for symptoms. Range is 0-70. Higher scores are worse.
Sexual function | Baseline
  Arizona Sexual Experiences Scale, adapted in terms of inclusive language. Range is 5-30. Higher scores are worse.
Sexual function | Week 4 of program
  Arizona Sexual Experiences Scale, adapted in terms of inclusive language. Range is 5-30. Higher scores are worse.
Sexual function | Week 8 of program
  Arizona Sexual Experiences Scale, adapted in terms of inclusive language. Range is 5-30. Higher scores are worse.
Sexual function | 3 months after the end of the program
  Arizona Sexual Experiences Scale, adapted in terms of inclusive language. Range is 5-30. Higher scores are worse.
Sexual function | 6 months after the end of the program
  Arizona Sexual Experiences Scale, adapted in terms of inclusive language. Range is 5-30. Higher scores are worse.
Alliance | Week 1 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 2 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 3 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 4 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 5 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 6 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 7 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Alliance | Week 8 of program
  Working Alliance with Therapist: Session Rating Scale. Four scales rated from 0-10 (range is 0-40), with higher scores indicating a better alliance.
Therapy group cohesion | Week 1 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 2 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 3 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 4 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 5 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 6 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 7 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.
Therapy group cohesion | Week 8 of program
  The Group Climate Questionnaire. 12 items total, 3 subscales. Items rated from 0 (not at all) to 7 (extremely). Range for each subscale due to averaging items is 0-7. Higher scores are better.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Pukall, PhD, Principal Investigator — Queen's University
Locations (1):
- Sexual Health Research Laboratory, Department of Psychology, Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to other researchers after publication of the results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be available to other researchers for 2 years after publication of the results.
Access Criteria: Please email the PI at caroline.pukall@queensu.ca